CLINICAL TRIAL: NCT03810001
Title: Use of Mechanical Stimulation to Active Oocytes Can Improve the Fertilization in Intracytoplasmic Sperm Injection Cycle
Brief Title: Mechanical Stimulation Improve the Fertilization in ICSI Cycle
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201801
Record Dates: First submitted 2019-01-07; First posted 2019-01-18 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Fertilization
Keywords: oocyte activation; intracytoplasmic sperm injection(ICSI); mechanical stimulation; 2PN rate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard ICSI procedure (No Intervention): a single spermatozoon was injected into the ooplasm
- modified ICSI procedure (Experimental): slight mechanical stimulation before standard ICSI procedure
  Interventions: Behavioral: Mechanical Stimulation

INTERVENTIONS:
Behavioral: Mechanical Stimulation — micromanipulation technique before insertion of the microinjection needle into the oocyte and expulsion of the spermatozoon
  Arms: modified ICSI procedure

SUMMARY:
Most fertilization failures after ICSI are caused by failure of oocyte activation defects. But, to date, there is no effective method to overcome this obstacle. To investigate the effect of mechanical stimulation on fertilization failures, investigators plan to recruit women undergoing ICSI treatment cycles. The retrieved sibling oocytes from the patients were randomly divided into two groups. The control group conducted the standard ICSI procedure, while the experimental group conducted the modified ICSI procedure.Consequently, the fertilization rate, 2PN (two pronuclei) rate, 1PN rate, oocyte degradation rate,and exploitable embryos on D3 were recorded to evaluate ICSI cycle outcomes.

DETAILED DESCRIPTION:
Normal fertilization is the critical for the success of ICSI. To investigate the effect of mechanical stimulation on fertilization, investigators plan to recruit women undergoing ICSI treatment cycles. Exclusion criteria: Patients older than 40 years, the maturation oocytes less than 6. The retrieved sibling oocytes from the patient were randomly divided into two groups. The control group conducted the standard ICSI procedure, while the experimental group conducted the modified ICSI procedure. The modified ICSI procedure involved a micromanipulation mechanical stimulation between insertion of the microinjection needle into the oocyte and expulsion of the spermatozoon from the needle to the ooplasm, without additional reagents treatment. Consequently, the fertilization rate, 2PN rate, 1PN rate, oocyte degradation rate, and exploitable embryos on D3 were recorded. The investigators aim to evaluate whether the mechanical stimulation can be used to improve the normal fertilization and embryo quality in ICSI cycles.

ELIGIBILITY:
Inclusion Criteria:

* oocytes number ≥ 8;
* women undergoing intracytoplasmic sperm injection cycle.

Exclusion Criteria:

* maturation oocytes number less than 6.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2019-11-20 (Estimated); Study Completion 2019-12-25 (Estimated)

PRIMARY OUTCOMES:
Normal fertilization rate | 6 months
  2PN (two pronuclei and two polar bodies) rate

SECONDARY OUTCOMES:
Feasibility and Efficacy of Mechanical Stimulation | 6 months
  Incidence of mechanical stimulation adverse events assessed by abnormally fertilization rate and oocytes degradation rate. Efficacy assessed by the exploitable embryo rate.

CONTACTS AND LOCATIONS:
Overall Officials: li bo, Study Chair — Reproductive Medicine Center, Tangdu Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China